CLINICAL TRIAL: NCT03168620
Title: Evaluation of the Effect of Glass Ionomer Cement as an Interim Restoration in Diagnosis of Pulpal Status in Permanent Teeth: A Prospective Randomized Clinical Trial
Brief Title: Effect of Glass Ionomer Cement as an Interim Restoration in Diagnosis of Pulpal Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Principal, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Monikakhokhar
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pulpitis
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITR group (Active Comparator): In ITR group after partial caries removal(PCR), interim therapeutic restoration of glass ionomer cement (GIC) Ketac molar was placed for one month before definitive adhesive restoration
  Interventions: Procedure: Restoration
- Non ITR group (Active Comparator): In NON-ITR group, cavity preparation was similar to ITR group, but definitive restoration was done in the same visit
  Interventions: Procedure: Restoration

INTERVENTIONS:
Procedure: Restoration
  Other Names: Filling

SUMMARY:
Aim: To evaluate whether glass ionomer interim therapeutic restoration (ITR) in asymptomatic teeth with deep cavities can help in determining the pulp status. Methodology: 146 mandibular molars with deep carious lesion having positive response to pulp sensitivity were randomly allocated to two study groups (75-ITR, 71- NON-ITR group). In the first group after partial caries removal(PCR), interim therapeutic restoration of glass ionomer cement (GIC) Ketac molar was placed for one month before definitive adhesive restoration. In NON-ITR group, cavity preparation was similar to ITR group, but definitive restoration was done in the same visit. Two examiners evaluated the clinical and radiographic outcomes for 18 months. Success was defined as absence of signs and symptoms of irreversible pulpitis and absence of periapical alterations.

DETAILED DESCRIPTION:
Introduction Preservation of pulp vitality while managing the deep carious lesions is often a great challenge and requires procedures like pulp capping and pulpotomy collectively termed as vital pulp therapy (VPT). Such treatment involves elimination of bacteria from pulp dentine complex and establishing an environment that will prevent any future bacterial contamination and improves survival prognosis. Management of deep carious lesions in recent years has changed from complete caries removal to partial caries removal. Partial caries removal has gained importance due to reduction in pulpal exposures, less postoperative complications, more preservation and maintenance of pulp tissue .

The important concern during VPT is accurate assessment of pulpal status. Methods to determine pulpal vitality include patient history, signs and symptoms, radiographs and pulp sensibility tests. One of the hallmarks of pulpal diagnosis is that it is difficult and has a high rate of inaccuracy. Pain on cold and hot stimuli cannot be considered as a reliable reference for making a treatment decision. Also insufficient evidence was found to determine the diagnostic accuracy of symptoms, signs, and diagnostic tests to assess the pulp status.

Studies using visual and histological inspection of exposed pulp to examine status of pulp reported marked variation in sensitivity of cold and electric pulp test from 0 .21 to 0.94, with relatively less variation in specificity from 0.73 to 0 .96.Sensitivity decreased to 67% when the spectrum of the disease was altered i.e. when asymptomatic teeth with deep carious lesions were included . Diagnosis of pulp status is often easy when there is a clear distinction between healthy and necrosed pulp however it is more difficult in asymptomatic teeth with deep carious lesions.

Recently, Coll et al. proposed that glass ionomer cement (GIC) as interim therapeutic restoration (ITR) improved pulpal diagnosis and VPT outcomes while interpreting diagnostic assessment based on clinical pulp therapy success. Vij et al. reported that GIC temporization for 1-3 months increased success of the subsequent VPT from 79% to 92% .However; both of the studies were retrospective and were in deciduous teeth.

No prospective clinical study has so far been conducted in permanent teeth that demonstrate the effectiveness of GIC and other adhesive restoration materials in determining the pulpal status. Aim of this double blinded randomized controlled trial was to assess the effectiveness of GIC interim restoration in determining the pulpal status of asymptomatic teeth with deep carious lesions. Null hypothesis was that GIC as ITR does not improve the clinician's diagnostic ability to determine the correct pulp clinical diagnosis and does not improve the treatment outcomes in vital pulp therapy.

Material and Methods:

Case Selection This prospective randomized clinical trial was conducted at the Department of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences, Rohtak, India. The study protocol was approved by the Ethical Committee (PGIDS/IEC/2015/64) of the Post Graduate Institute of Dental Sciences. A total of 146 patients were included with an age range of 15-54 years. The inclusion criteria for the study were: 1) mature permanent mandibular molars having deep carious lesions involving half or more of the dentine detected by radiographic examination, 2) pulp sensibility confirmed using the electric pulp test (Digitest D626D; Parkell Electronics, New York, NY) and the cold test (Endo frost, Coltene, Whaledent), 3) absence of apical and furcal radiolucency determined by radiographic examination, 4) absence of clinical symptoms of irreversible symptoms, fistula, swelling and abnormal tooth mobility. Clinical diagnosis of vital pulp was made by the chief supervisor (Sanjay Tewari) on the basis of radiographic and clinical examination and the pulp sensibility tests. Patients were excluded if they presented with signs and symptoms of irreversible pulpitis, had negative response to vitality tests before or after ITR, diabetic, immunocompromised, pregnant, or had a positive history of antibiotic use in past one month or required antibiotic prophylaxis. Informed consent explaining benefits and risks of treatment was taken from patients before participation in the trial.

Sample Size Calculation and Randomization The sample size calculation was done on the basis of difference in the percentage of success of vital pulp therapy using GIC (98%) versus non-GIC group (75%) (12) α=5% with a power of 90%. This indicated the need for 48 restorations per treatment group. Given an expected attrition rate of 20%, 60 teeth were included in each treatment group. Randomization was developed to eliminate any bias on the part of the investigators and to equalize the number of patients between the 2 treatment groups. Using an equal proportion randomization allocation ratio, one of the investigators (M.J) created envelopes containing concealed assignment codes that were assigned sequentially to eligible patients.

Clinical Procedure The procedure was performed under local anesthesia and rubber dam isolation. Carious tissue from the lateral walls and dentinoenamel junction was removed completely by using low-speed metal burs and/or hand excavator. Superficial necrotic dentin was removed from the pulpal and axial wall using low speed round bur. A layer of soft, wet carious dentin was left adjacent to pulpal wall. The cavity was cleaned with distilled water and dried with sterile filter paper. In group ITR, the cavity was filled with GIC ( Ketac Molar (3M ESPE, St. Paul, Minn., USA).Cavity was reopened after 1 months in asymptomatic patients , restoration was removed completely ,base of resin modified glass ionomer cement(RMGIC) (Fuji Lining LC;GC,Tokyo,Japan)was applied and cavity was restored with resin composite(Tetric N-Ceram;Ivoclar Vivadent) according to manufacturer instructions.

In NON-ITR group, cavity preparation was done similar to ITR group, after partial caries excavation ,base of RMGIC (Fuji Lining LC;GC,Tokyo,Japan) was applied and all cavities were restored with resin composite(Tetric N-Ceram;Ivoclar Vivadent) according to manufacturer instructions.

Outcome Assessment Two blinded examiners assessed the clinical and radiographic outcomes of test and control treatments at 1, 3, 6, 12, 18 months after treatment. Success was defined as absence of signs and symptoms of irreversible pulpitis (spontaneous pain, fistula and swelling), positive response to pulp sensibility tests and absence of periapical alterations (radiolucency at furcal or periapical region, calcification) (combined outcome). Pretreatment pulpal diagnosis was considered successful when teeth treated with or without ITR were diagnosed as vital and none of clinical and radiographic signs and symptoms of failure developed during 18 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* mature permanent mandibular molars having deep carious lesions involving half or more of the dentine detected by radiographic examination,
* pulp sensibility confirmed using the electric pulp test (Digitest D626D; Parkell Electronics, New York, NY) and the cold test (Endo frost, Coltene, Whaledent),
* absence of apical and furcal radiolucency determined by radiographic examination,
* absence of clinical symptoms of irreversible symptoms, fistula, swelling and abnormal tooth mobility.
* Clinical diagnosis of vital pulp was made on the basis of radiographic and clinical examination and the pulp sensibility tests.

Exclusion Criteria:• if they presented with signs and symptoms of irreversible pulpitis,

* had negative response to vitality tests before or after ITR,
* diabetic, immunocompromised,
* pregnant,
* had a positive history of antibiotic use in past one month or required antibiotic prophylaxis.

Ages: 15 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
clinical success | 18 months
  Success was defined as absence of signs and symptoms of irreversible pulpitis (spontaneous pain, fistula and swelling), positive response to pulp sensibility tests.
radiographic success | 18 months
  Absence of periapical alterations (radiolucency at furcal or periapical region, calcification). Pretreatment pulpal diagnosis was considered successful when teeth treated with or without ITR were diagnosed as vital and radiographic signs and symptoms of failure developed.

IPD SHARING:
Plan to Share IPD: Yes